CLINICAL TRIAL: NCT04805190
Title: Neural Mechanisms Underlying Psychosocial Contributions to Ethnic Group Differences in Pain
Brief Title: Study of Pain Catastrophizing-2 (SPAC-2)
Acronym: SPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB202100297 -N; K22NS102334 (NIH); OCR40441 (Other: UF OnCore)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
Keywords: catastrophizing; cognitive-behavior therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a single session cognitive-behavioral intervention to reduce pain catastrophizing or a pain education control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Catastrophizing Reduction Group (Experimental): This group will be assigned to a 30-minute, single-session cognitive-behavioral intervention designed to reduce pain catastrophizing.
  Interventions: Behavioral: Cognitive-Behavioral Intervention
- Pain Education Group (Active Comparator): This group will receive general information about the neurobiology of pain and knee OA.
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention — This intervention comprises three components: 1) general education about pain (e.g., pain pathways) and a rationale for the intervention (e.g., gate control theory); 2) impact of positive and negative pain-related thoughts on neural process of pain; and 3) a guided imaginal pain exposure exercise.
  Arms: Pain Catastrophizing Reduction Group
Behavioral: Pain Education — General information about the neurobiology of pain and knee osteoarthritis will be given to participants assigned to this intervention.
  Arms: Pain Education Group

SUMMARY:
This study experimentally manipulates pain catastrophizing in order to investigate the neural mechanisms by which pain catastrophizing influences the experience of pain in different ethnic groups among adults with knee osteoarthritis. Participants will be randomized to either a single session cognitive-behavioral intervention to reduce pain catastrophizing or a pain education control group.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA

Exclusion Criteria:

* Younger than 45 years of age or older than 85 years of age
* Prosthetic knee replacement or other clinically significant surgery to the arthritic knee
* Uncontrolled hypertension (>150/95)
* Heart disease including heart failure
* Peripheral neuropathy in which pain testing was contraindicated
* Systemic rheumatic disorders including rheumatoid arthritis, systemic lupus erythematosus, gout, and fibromyalgia
* Neurological diseases such as Parkinson's, multiple sclerosis, stroke with loss of sensory or motor function, or uncontrolled seizures
* Significantly greater pain in body sites other than in the knee
* Daily opioid use
* Hospitalization within the preceding year for psychiatric illness
* Currently pregnant or nursing/breastfeeding

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Catastrophizing Scale (PCS) | Baseline; Day 2
  13-item scale that assesses catastrophic thinking associated with pain. The study team will administer the PCS using traditional instructions (a measure of trait catastrophizing) and instructions to assess situation-specific catastrophizing ("Thinking back to your experience during the laboratory pain testing"). Thoughts and feelings concerning pain are ranked on a 0-4 scale, with 0 being the patient has this thought/feeling 'not at all' to 4, the patient has this thought feeling 'all the time.'

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Terry, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No